CLINICAL TRIAL: NCT07031323
Title: OnTrackCF: Engagement, Feasibility, and Acceptability Study
Acronym: OnTrackCF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Johns Hopkins University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gregory Sawicki, Co-Chair of the Success with Therapies Research Consortium, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00050537
Record Dates: First submitted 2025-06-09; First posted 2025-06-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis (CF); Cystic Fibrosis - Complete
Keywords: adherence; mHealth; mobile health; digital health; medication adherence; CFTR Modulators
MeSH Terms: conditions — Cystic Fibrosis; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participation (Experimental): Participants eligible to enroll will be provided with the OnTrackCF app (intervention), and will use the app for 4-12 weeks before completing feasibility measures and a qualitative interview.
  Interventions: Behavioral: OnTrackCF

INTERVENTIONS:
Behavioral: OnTrackCF — OnTrackCF is a mHealth application co-developed with Upstream Dream. It is designed specifically to track and support adherence to CFTR modulator therapy. The app allows users to track their modulator intake and disease symptoms while supporting their adherence goals using Behavioral Change Techniques (BCTs) with empirical evidence of efficacy. The BCTs are administered primarily in the form of messages designed to deliver specific BCTs. The app sends up to 3 adherence support messages per day and provides detailed data to the user about their adherence levels, adherence goals, and disease symptoms. This process will continue until we reach an N=60 AWCF enrolled OR demonstrate that we have achieved 12 weeks of sustained user engagement with the app.

SUMMARY:
This is a multi-site, nonrandomized study using mixed methods approach to evaluate the feasibility, acceptability, and user engagement of OnTrackCF for adults with Cystic Fibrosis (AWCF).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with CF
2. 18+ years of age
3. Prescribed a CFTR modulator therapy to be taken twice a day
4. Can speak and read English
5. Have regular access to an iOS or Android tablet or smartphone with internet access.

Exclusion Criteria:

1) Any situation, in the opinion of the Investigator, that would compromise the safety of the patient or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
System Usability Survey (SUS) | through study completion, projected to be 1 year
  By the last round of testing, the System Usability Survey (SUS) will have a median score of 75%.
Intervention Feasibility and Acceptability (iFAQ) | through study completion, projected to be 1 year
  By the last round of testing, the Intervention Feasibility and Acceptability (iFAQ) OnTrackCF scales (Engagement, Feasibility, Acceptability, Usefulness, and Satisfaction) will each have a median score of ≥4 (out of 5).

SECONDARY OUTCOMES:
Onboarding Completion | through study completion, projected to be 1 year
  By the last round of testing, 90% of participants will complete the app onboarding process.
Engagement with app features | through study completion, projected to be 1 year
  By the last round of testing, 70% of onboarded participants will engage with at least one app feature at least once during each week of their study period.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Riekert, PhD, Principal Investigator — Johns Hopkins University; Gabriela Oates, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided